CLINICAL TRIAL: NCT07389759
Title: Impact of CADx on Endoscopists' Histologic Characterization of Diminutive Colorectal Polyps
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Xiaobo Li, Chief physician, Shanghai Jiao Tong University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: KY2024-080-A-02
Record Dates: First submitted 2026-01-29; First posted 2026-02-05 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-01

CONDITIONS: Colorectal Polyps

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Standard Colonoscopy (No CADx Assistance) (No Intervention): Endoscopists perform optical diagnosis of diminutive colorectal polyps (≤5 mm) during colonoscopy using narrow-band imaging (NBI) without any CADx assistance.
- CADx Without Predicted Probability (Experimental): Endoscopists perform optical diagnosis of diminutive colorectal polyps (≤5 mm) during colonoscopy using NBI, with CADx-displayed NICE classification predictions but without any predicted probability information.
  Interventions: Device: CADx-Assisted Endoscopic Diagnosis System Without Predicted Probability Display
- CADx With PPredicted Probability (Experimental): Endoscopists perform optical diagnosis of diminutive colorectal polyps (≤5 mm) during colonoscopy using NBI, with CADx-displayed NICE classification predictions and accompanying predicted probability information.
  Interventions: Device: CADx-Assisted Endoscopic Diagnosis System With Predicted Probability Display

INTERVENTIONS:
Device: CADx-Assisted Endoscopic Diagnosis System Without Predicted Probability Display — CADx-assisted optical diagnosis (NBI; predicted probability not displayed). Endoscopists perform optical diagnosis of diminutive colorectal polyps (≤5 mm) during colonoscopy using narrow-band imaging (NBI) with CADx-displayed NICE classification predictions for each polyp. In this arm, the CADx output is displayed without any predicted probability information.
  Arms: CADx Without Predicted Probability
Device: CADx-Assisted Endoscopic Diagnosis System With Predicted Probability Display — CADx-assisted optical diagnosis (NBI; predicted probability displayed). Endoscopists perform optical diagnosis of diminutive colorectal polyps (≤5 mm) during colonoscopy using narrow-band imaging (NBI) with CADx-displayed NICE classification predictions for each polyp. In this arm, the CADx output is displayed with accompanying predicted probability information.
  Arms: CADx With PPredicted Probability

SUMMARY:
This study evaluates the impact of CADx assistance on endoscopists' histologic characterization of diminutive colorectal polyps (≤5 mm) during colonoscopy. The primary objective is to determine whether CADx assistance increases the proportion of endoscopists who meet PIVI-related performance thresholds, thereby supporting implementation of the "resect and discard" and "diagnose and leave" strategies in routine clinical practice.

DETAILED DESCRIPTION:
This study evaluates the impact of CADx assistance on endoscopists' histologic characterization of diminutive colorectal polyps (≤5 mm) during colonoscopy. The primary objective is to determine whether CADx assistance increases the proportion of endoscopists who meet PIVI-related performance thresholds, thereby supporting implementation of the "resect and discard" and "diagnose and leave" strategies in routine clinical practice.

In this randomized controlled trial, endoscopists will be assigned to one of three arms: no CADx assistance, CADx assistance without predicted probability, or CADx assistance with predicted probability. The CADx system provides NICE-based histology predictions (Type 1 vs Type 2), which endoscopists may use to support optical diagnosis and subsequent management decisions, including surveillance interval recommendations when applicable. Outcomes will compare endoscopist-level pass rates and diagnostic performance metrics relevant to PIVI-based adoption, with histopathology as the reference standard where applicable.

ELIGIBILITY:
Inclusion Criteria:

* Endoscopists with NBI experience

Exclusion Criteria:

-Endoscopists without colonoscopy and NBI experience

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 363 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Pass rate for the "resect and discard" strategy | 14 days
  Proportion of endoscopists who achieve ≥90% accuracy in correctly predicting the patient's recommended surveillance colonoscopy interval according to the 2020 U.S. Multi-Society Task Force (USMSTF) consensus recommendations.
Pass rate for the "diagnose and leave" strategy | 14 days
  Proportion of endoscopists who achieve a negative predictive value (NPV) ≥90% for neoplastic lesions among rectosigmoid polyps, when predictions are made with high diagnostic confidence

SECONDARY OUTCOMES:
Pass rate for the ESGE 2020-based "resect and discard" strategy | 14 days
  The proportion of endoscopists who achieve at least 90% accuracy in correctly predicting the patient's recommended next surveillance colonoscopy interval, using surveillance recommendations based on the ESGE 2020 guideline.
Pass rate for the APWG 2022-based "resect and discard" strategy | 14 days
  The proportion of endoscopists who achieve at least 90% accuracy in correctly predicting the patient's recommended next surveillance colonoscopy interval, using surveillance recommendations based on the APWG 2022 consensus.
Pass rate for the China 2023-based "resect and discard" strategy | 14 days
  The proportion of endoscopists who achieve at least 90% accuracy in correctly predicting the patient's recommended next surveillance colonoscopy interval, using surveillance recommendations based on the Chinese 2023 consensus.
SODA-1 achievement rate | 14 days
  The proportion of endoscopists who, when reporting high diagnostic confidence, meet the SODA-1 performance thresholds for diagnosing neoplastic pathology in diminutive rectosigmoid polyps, as assessed by sensitivity of at least 90% and specificity of at least 80%, with histopathology as the reference standard.
SODA-2 achievement rate | 14 days
  The proportion of endoscopists who, when reporting high diagnostic confidence, meet the SODA-2 performance thresholds for diagnosing neoplastic pathology in diminutive colorectal polyps, as assessed by sensitivity of at least 80% and specificity of at least 80%, with histopathology as the reference standard.
Proportion of high-confidence optical diagnoses | 14 days
  For each endoscopist, the percentage of polyp assessments that are labeled as high diagnostic confidence among all polyp assessments performed.
Accuracy of high-confidence optical diagnosis (neoplastic vs non-neoplastic) | 14 days
  For each endoscopist, the percentage of correct classifications (neoplastic vs non-neoplastic) among assessments labeled as high diagnostic confidence, using histopathology as the reference standard.

IPD SHARING:
Plan to Share IPD: No